CLINICAL TRIAL: NCT00949988
Title: A Phase I/II Study of Dasatinib and Rituximab for Relapsed/Refractory Chronic Lymphocytic Leukemia
Brief Title: A Study of Dasatinib and Rituximab for Relapsed/Refractory Chronic Lymphocytic Leukemia
Acronym: BMS-CA180105
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Three subjects were enrolled and all three subjects withdrew.
Sponsor: University of California, San Diego (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Thomas Kipps, Professor, University of California, San Diego
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCSD 110054 - Prev 080422
Record Dates: First submitted 2009-07-28; First posted 2009-07-31 (Estimated); Results first posted 2019-08-14 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-07

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Chronic Lymphocytic Leukemia; CLL; Dasatinib; Rituximab; Relapsed; Refractory
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Recurrence | interventions — Dasatinib; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dasatinib - 100 mg (Phase I) (Active Comparator): Dasatinib - 100 mg (Phase I)
  Interventions: Drug: Dasatinib and Rituximab
- Dasatinib - 70 mg (Phase I) (Active Comparator): Dasatinib - 70 mg (Phase I)
  Interventions: Drug: Dasatinib and Rituximab

INTERVENTIONS:
Drug: Dasatinib and Rituximab — In Phase I, subjects will be enrolled into a "3+3" dose escalation scheme with two dasatinib cohort doses of 70 mg QD and 100 mg QD to be given continuously during each 28-day cycle. All subjects will also receive rituximab 500 mg/m2 on day 1 of each cycle (375 mg/m2 on day 1 of cycle 1 only). There will be a pre-phase for each dose cohort when subjects will receive single-agent dasatinib from days -7 to -1 to allow for PK and PD assessment. Cohorts will be assessed for dose-limiting toxicities for two cycles before accrual of additional

SUMMARY:
This is an open-label phase I/II study that will investigate the combination of dasatinib and rituximab therapy in patients with relapsed/refractory CLL. In phase I, eligible subjects will take either 100 mg or 140 mg of dasatinib daily along with rituximab on day 1 of each cycle for 6 cycles. In phase II, eligible subjects will all receive the same dose of dasatinib, as established in the phase I portion, along with rituximab on day 1 of each cycle for 6 cycles.

The investigators hypothesize that the combination of dasatinib and rituximab will demonstrate efficacy in the treatment of patients with relapsed/refractory CLL.

DETAILED DESCRIPTION:
In phase I, patients will be enrolled in a standard "3+3" dose escalation scheme with two dasatinib cohort doses of 100 mg QD and 140 mg QD x 28 days/cycle with rituximab 500 mg/m2 on day 1 of each cycle (375 mg/m2 on day 1 of cycle 1 only). During the first cycle of each dose cohort patients will receive dasatinib on days -7 to 0 to allow for pharmacokinetic and pharmacodynamic analysis of single agent dasatinib dosing. Cohorts will be assessed for DLTs during the first 2 cycles. Treatment will continue for 6 cycles or until intolerable toxicity or disease progression. It is estimated that accrual of 3-6 patients will be completed in 4-6 months depending on DLTs observed.

The dasatinib dose established in phase I will move forward to the phase II setting. If there are no DLTs, the phase II dose will be chosen based on PD parameters. Dasatinib will be administered for 28 days/cycle with rituximab 500 mg/m2 on day 1 of each cycle (375 mg/m2 on day 1 of cycle 1 only) for 6 cycles or until intolerable toxicity or disease progression. For this portion of the study, up to an additional 22 patients will be enrolled over a 6-month period for a total of 28 patients at the chosen dose level.

For both, phase I and II, patients will complete up to six cycles of D+R therapy and endpoints will be evaluated 8 weeks after treatment. Patients will be followed until disease progression, study withdrawal or death. Patients with a PR or CR will be eligible to remain on dasatinib alone.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Confirmed immunohistological diagnosis of B-cell CLL and Rai Stage III or IV disease, or stage 0-II disease that meets NCIWG criteria for active disease as indicated by any one of the following disease-related symptoms:

   * Weight loss ≥ 10% within the previous 6 months
   * Extreme fatigue
   * Fever greater than 100.5 degrees Fahrenheit for ≥ 2 weeks without evidence of infection
   * Night sweats without evidence of infection
   * Evidence of progressive marrow failure based on the development or worsening of anemia (< 10 g/dL) or thrombocytopenia (< 100,000 cells/mL)
   * Autoimmune anemia and/or thrombocytopenia poorly responsive to corticosteroid therapy
   * Massive (> 6 cm below the left costal margin) or progressive splenomegaly
   * Bulky (>10 cm in cluster) or progressive lymphadenopathy
   * Progressive lymphocytosis with > 50% increase over a 2-month period, or anticipated doubling time < 6 months
2. Relapsed/ Refractory CLL that has progress with ≥1 prior treatment including a purine nucleoside analog-containing regimen, alkylating agent, or antibody (rituximab or alemtuzumab) or intolerance to purine nucleoside analog-containing therapy or unwilling to receive chemotherapy treatment.
3. Age 18 or older
4. ECOG Performance Status 0-2 (Appendix B)
5. Adequate organ function:

   * Serum creatinine < 2x the institutional upper limit of normal (ULN)
   * Total bilirubin < 2x the institutional ULN
   * AST, ALT < 2.5x the institutional ULN
   * Serum sodium, potassium, magnesium, phosphate and calcium > the institutional lower limit of normal (LLN)
6. Ability to take oral medication (dasatinib must be swallowed whole)
7. Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (sensitivity ≤ 25 IU/L HCG) within 72 hrs prior to the start of study drug administration
8. Persons of reproductive potential must agree to use an adequate method of contraception throughout treatment and for at least 4 weeks after study drug is stopped
9. Ability to understand and the willingness to sign a written informed consent document

EXCLUSION CRITERIA:

1. No prior CLL-related treatment within 28 days before starting treatment with dasatinib.
2. No concurrent use of other investigation agent.
3. Concurrent medical condition which may increase the risk of toxicity, including:

   * Uncontrolled or significant cardiovascular disease, including:

     * Myocardial infarction, congestive heart failure or uncontrolled angina within 6 months
     * Diagnosed congenital long QT syndrome
     * Any history of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or Torsade de Pointes)
     * Prolonged QTcF interval on pre-entry ECG (> 450 msec)
     * 2nd/3rd degree heart block, uncontrolled hypertension or heart rate < 50
   * History of significant bleeding disorder unrelated to CLL, including:

     * Diagnosed congenital bleeding disorder (e.g., von Willebrand's disease)
     * Diagnosed acquired bleeding disorder within one year (e.g., acquired anti-factor VIII antibodies)
     * Ongoing or recent significant GI bleeding within 3 months
   * Hypokalemia or hypomagnesemia if it cannot be corrected
   * Pleural or pericardial effusion of any grade
   * Past or current malignancy, except for:

     * Cervical carcinoma Stage 1B or less
     * Non-invasive basal cell and squamous cell skin carcinoma
     * Malignant melanoma with a complete response of a duration of > 10 years
     * Other cancer diagnoses with a complete response of a duration of > 5 years
   * Major systemic or other illness including active infection or active secondary malignancy that would, in the opinion of the Investigator, interfere with the patient's ability to comply with the protocol, compromise patient safety, or interfere with the interpretation of the study results
4. No history of allergic reaction to dasatinib.
5. Use of Prohibited Concomitant Medications

   Subjects requiring any of the following prohibited therapies should not be enrolled:
   * Bisphosphonates Intravenous bisphosphonates will be withheld for the first 8 weeks of treatment due to the risk of hypocalcemia. After the need for Ca2+ supplementation has been assessed and levels documented to be >LLN, subjects on prior bisphosphonate may be restarted with caution at the Investigator's discretion.
   * CYP3A4 Inhibitors/Inducers/Substrates Dasatinib is primarily metabolized by the CYP3A4 enzyme. Therefore, potent inhibitors of CYP3A4 are prohibited during study; for such medications, a wash-out period of ≥ 7 days is required prior to starting dasatinib. Subjects should be advised not to consume substantial quantities of grapefruit juice.
   * Drugs that may increase dasatinib plasma concentrations:

   CYP3A4 Inhibitors: Dasatinib is a CYP3A4 substrate. Concomitant use of dasatinib and drugs that inhibit CYP3A4 (e.g., ketoconazole, itraconazole, erythromycin, clarithromycin, ritonavir, atazanavir, indinavir, nefazodone, nelfinavir, saquinavir, telithromycin) may increase exposure to dasatinib and should be avoided.

   In patients receiving treatment with dasatinib, close monitoring for toxicity and a dasatinib dose reduction should be considered if systemic administration of a potent CYP3A4 inhibitor cannot be avoided.

   -Drugs that may decrease dasatinib plasma concentration: CYP3A4 Inducers: Drugs that induce CYP3A4 activity may decrease dasatinib plasma concentrations. In patients in whom CYP3A4 inducers (eg, dexamethasone, phenytoin, carbamazepine, rifampicin, phenobarbital) are indicated, alternative agents with less enzyme induction potential should be used. If dasatinib must be administered with a CYP3A4 inducer, a dose increase in dasatinib should be considered and approved by the principal investigator.

   -Drugs that may have their plasma concentration altered by dasatinib: CYP3A4 Substrates: CYP3A4 substrates known to have a narrow therapeutic index such as alfentanil, astemizole, terfenadine, cisapride, cyclosporine, fentanyl, pimozide, quinidine, sirolimus, tacrolimus, or ergot alkaloids (ergotamine, dihydroergotamine) should be administered with caution in patients receiving dasatinib.
   * Less-potent inhibitors, inducers, and substrates of CYP3A4 are restricted.
   * St. John's Wort (Hypericum perforatum):

   May decrease dasatinib plasma concentrations unpredictably. Patients receiving dasatinib should not take St. John's wort.
   * Antacids Nonclinical data demonstrate that the solubility of dasatinib is pH dependent. Simultaneous administration of dasatinib with antacids should be avoided. If antacid therapy is needed, the antacid dose should be administered at least 2 hours prior to or 2 hours after the dose of dasatinib.
   * H2 Blockers/Proton Pump Inhibitors Long-term suppression of gastric acid secretion by H2 blockers or proton pump inhibitors (eg, famotidine and omeprazole) is likely to reduce dasatinib exposure. The concomitant use of H2 blockers or proton pump inhibitors with dasatinib is not recommended. The use of antacids should be considered in place of H2 blockers or proton pump inhibitors in patients receiving dasatinib therapy.
   * Medications that prolong QT Interval

   Subjects enrolled in this study should not take or begin to take concomitant medications known to prolong the QT interval. If such medications are already being taken by the patient before study starts, a wash-out period of ≥ 7days is required prior to starting dasatinib. Medications known to prolong the QT interval and/or are generally accepted to have a risk of causing Torsades de Pointes ventricular arrhythmia are (see http://www.qtdrugs.org/medical-pros/drug-lists/drug-lists.htm):
   * Quinidine, procainamide, disopyramide
   * Amiodarone, sotalol, ibutilide, dofetilide
   * Erythromycin, clarithromycin
   * Chlorpromazine, haloperidol, mesoridazine, thioridazine, pimozide
   * Cisapride, bepridil, droperidol, methadone, arsenic, chloroquine, domperidone, halofantrine, levomethadyl, pentamidine, sparfloxacin, lidoflazine Should the Investigator believe that beginning therapy with a potentially QT prolonging medication (other than the ones explicitly prohibited) is vital to an individual subject's care, the Investigator must check that the subject's prior on-therapy ECG has not shown a QTcF ≥ 450 msec or an increase in QTc ≥ 60 msec over the baseline value.

     * Anticoagulants and Medications that inhibit Platelet Function Caution should be exercised if patients are required to take medications that inhibit platelet function or anticoagulants.

   Subjects enrolled in this study should not take concomitant medications that durably inhibit platelet function. For such medications, a wash-out period of ≥ 7days is required prior to starting dasatinib. (Agents that inhibit platelet function transiently or inhibit coagulation by other mechanisms are restricted.)

   Medications that directly and durably inhibit platelet function include:
   * aspirin or aspirin-containing combinations, clopidogrel, dipyridamole
   * tirofiban, dipyridamole, epoprostenol, eptifibatide, cilostazol, abciximab, ticlopidine, cilostazol

   Medications that directly and durably inhibit anticoagulation include:
   * warfarin, heparin/low molecular weight heparin [e.g., danaparoid, dalteparin, tinzaparin, enoxaparin]
   * Exceptions: low-dose warfarin for prophylaxis to prevent catheter thrombosis, and heparin for flushes of IV lines.
6. Women who are pregnant (including having a positive pregnancy test) or breastfeeding, or unable/unwilling to practice an acceptable method to avoid pregnancy for the entire study period and for at least 4 weeks after cessation of study drug, or men who are sexual partners thereof.

   * Sexually active women of childbearing potential (WOCBP) must use an effective method of birth control during the course of the study, in a manner such that risk of failure is minimized. Prior to study enrollment, WOCBP must be advised of the importance of avoiding pregnancy during trial participation and the potential risk factors for an unintentional pregnancy.
   * All WOCBP MUST have a negative pregnancy test prior to first receiving dasatinib. If the pregnancy test is positive, the patient must not receive dasatinib and must not be enrolled in the study.
7. Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (e.g., infectious) illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2009-05 (Actual); Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Januario Castro, M.D., Principal Investigator — Clinical Professor, Blood and Bone Marrow Transplant Division; Thomas J Kipps, M.D., Ph.D., Principal Investigator — Professor of Medicine, Evelyn and Edwin Tasch Chair in Cancer Research in the UCSD School of Medicine
Locations (1):
- University of California San Diego Moores Cancer Center, La Jolla, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: This study only enrolled three subjects and all three subjects withdrew before study completion.
Period: Overall Study
Arm/Group | All Participants
Started | 3
Completed | 0
Not Completed | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: Phase I: To Determine the Dose-limiting Toxicities (DLTs) and Maximum Tolerated Dose (MTD) of D+R Therapy in Patients With Relapsed/Refractory CLL
Time Frame: 1 year
Population: This study only enrolled three participants and all three participants withdrew. No data analysis was performed.
Arm/Group | All Participants
Number analyzed (Participants) | 0

2. Secondary Outcome: To Assess the Safety Profile of D+R in Relapsed/Refractory CLL Patients
Time Frame: 2 years
Population: This study only enrolled three participants and all three participants withdrew. No data analysis was performed.
Arm/Group | All Participants
Number analyzed (Participants) | 0

3. Secondary Outcome: To Assess Duration of Progression-free Survival
Time Frame: 5 years
Population: This study only enrolled three participants and all three participants withdrew. No data analysis was performed.
Arm/Group | All Participants
Number analyzed (Participants) | 0

4. Secondary Outcome: To Assess Minimal Residual Disease (MRD) by Flow Cytometry
Time Frame: 2 years
Population: This study only enrolled three participants and all three participants withdrew. No data analysis was performed.
Arm/Group | All Participants
Number analyzed (Participants) | 0

5. Secondary Outcome: To Determine the Effect of Several Prognostic Factors Including CD38 Expression, ZAP-70 Expression, Immunoglobulin Variable Heavy Chain (VH) Gene Mutation Status and Cytogenetic/FISH Profile on Treatment Response.
Time Frame: 2 years
Population: This study only enrolled three participants and all three participants withdrew. No data analysis was performed.
Arm/Group | All Participants
Number analyzed (Participants) | 0

6. Secondary Outcome: To Evaluate in CLL Cells Pharmacodynamic (PD) Parameters Including the Following: in Vivo Signal Transduction Events, Levels of Cellular Apoptosis and Regulation of Apoptosis Related Genes and Proteins.
Time Frame: 2 years
Population: This study only enrolled three participants and all three participants withdrew. No data analysis was performed.
Arm/Group | All Participants
Number analyzed (Participants) | 0

7. Secondary Outcome: To Evaluate Pharmacokinetics for Dasatinib in the Treated Patients
Time Frame: 2 years
Population: This study only enrolled three participants and all three participants withdrew. No data analysis was performed.
Arm/Group | All Participants
Number analyzed (Participants) | 0

8. Secondary Outcome: A Multi-Center Phase I/II Study of Dasatinib and Rituximab for Relapsed/Refractory Chronic Lymphocytic Leukemia
Description: Phase II:
  To determine the efficacy of D+R treatment in patients with relapsed/refractory CLL as measured by complete and partial response rates
Time Frame: 2 years
Population: This study only enrolled three participants and all three participants withdrew. No data analysis was performed.
Arm/Group | All Participants
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 3/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=3)
Rigors (General disorders) | 1 (1)
Sialoadenitis (Ear and labyrinth disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes